CLINICAL TRIAL: NCT07332104
Title: The Application of Extracellular Vesicle Detection in Gastric Juice Based on Metamaterial Sensing in the Diagnosis of Gastric Cancer and Related Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Min Li, Professor, Beijing Friendship Hospital
Other Study IDs: BFHZS20240020; No. BFHZS20240020 (Other Grant/Funding Number: the Ethics Committee of Beijing Friendship Hospital, Capital Medical University)
Record Dates: First submitted 2025-12-14; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer (GC); Gastric Cancer (Diagnosis)
Keywords: Gastric cancer; Extracellular vesicles
MeSH Terms: conditions — Stomach Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Extracellular vesicles
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- gastric cancer: Patients diagnosed with gastric cancer
  Interventions: Diagnostic Test: In vitro surface plasmon resonance detection

INTERVENTIONS:
Diagnostic Test: In vitro surface plasmon resonance detection — Gastric juice from patients was removed for isolation of extracellular vesicles and surface plasmon resonance detection in vitro

SUMMARY:
After obtaining informed consent from the patients, all the medical history and treatment records of the patients who underwent gastroscopy since the onset of the disease, as well as gastric fluid samples, including laboratory and imaging data, were collected and recorded. The medical history and treatment records and gastric fluid samples were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent gastroscopy and treatment at the Endoscopy Center of Beijing Friendship Hospital, Capital Medical University, and received pathological biopsy.
* Previous gastroscopy suggested the possibility of lesions.
* No previous history of gastrointestinal cancer.

Exclusion Criteria:

* Patients could not cooperate with the examination or had contraindications to endoscopy.
* Previous history of gastrointestinal tumors, gastrointestinal surgery, physical and chemical injuries of the gastrointestinal tract.
* Severe bile reflux.
* Take simethicone and other defoaming agents before examination.
* Patients with serious diseases of heart, lung, kidney, brain, blood and other important organs.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gastric cancer and non-cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Surface plasmon resonance(SPR) detection of extracellular vesicles in gastric juice of patients with gastric cancer has large shift and spectral changes | baseline

DOCUMENTS (2):
  • Study Protocol (2025-12-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT07332104/Prot_000.pdf
  • Informed Consent Form (2025-12-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT07332104/ICF_001.pdf